CLINICAL TRIAL: NCT04102384
Title: Usability and Satisfaction With an Electronic Survey Administration Application in General Population
Acronym: CePRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Cenduit LLC (Industry)
Responsible Party: Principal Investigator, Ramya Sita Palacholla, MD, MPH, Partners Healthcare, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019P002811
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Surveys; Usability; Healthy
Keywords: Electronic Patient Reported Outcomes

STUDY DESIGN:
Intervention Model Description: Intervention- one group will use a smartphone application to fill out surveys while the other group fills out surveys via an emailed embedded link.
Who Masked: Participant
Masking Description: Participants will not know which group (smart phone or embedded link) is the intervention vs. control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants will be enrolled for a period of 4 weeks. At baseline, we will collect demographic information on participants. During the study, participants will be asked to fill out daily and weekly surveys using an electronically link sent via email. Additionally, participants will be asked to fill out one survey once a week during the study period.
- Intervention Group (Experimental): Participants will be enrolled for a period of 4 weeks. At baseline, we will collect demographic information on participants. During the study, participants will be asked to fill out daily and weekly surveys using the e-PRO app. Additionally, participants will be asked to fill out one survey once a week during the study period. A subgroup of these participants will be asked to complete an additional interview to collect more information on their experiences using the mobile app.
  Interventions: Other: e-PRO App

INTERVENTIONS:
Other: e-PRO App — The e-PRO app is designed to further facilitate the delivery of PRO instruments in a convenient manner to participants. Through its computing capability, and user-friendly interface, the e-PRO app can collect data and implement complex scoring requirements, thus supporting the delivery of self-administered survey questionnaires.
  Arms: Intervention Group

SUMMARY:
The goal of the study is to assess the usability and satisfaction of an electronic patient reported outcomes (e-PRO) mobile application. The secondary aim is to assess and compare response rates between two study groups (e-PRO group vs REDCap survey group). A potential differentiating factor between delivering surveys via smart phone and other electronic modes of delivery is the perceived advantage of being able to conveniently complete survey questionnaires at any time and any location. This could help address certain limitations of the quantitative survey method such as recall bias. Furthermore, the portability, connectivity and ubiquity of smartphones may reduce the amount of training or instructions required for users to complete a survey questionnaire on a smartphone.

DETAILED DESCRIPTION:
Patient-reported outcomes (PROs) are vital to understanding the impact of a medical condition and treatment from the participant's perspective. However, the collection of data can be inconsistent in both administration and completion due to the method of delivery. Thus, careful consideration of the data collection mode is needed to ensure the quality of the data. The method of delivery has been shown to have a direct effect on the survey response rates thereby ensuring the validity of the data analyses and results. Previous studies have demonstrated an increase in Web-based survey response rates as compared to paper-based survey response rates. Novel methods of collecting PROs may help to streamline both the process and collection of PROs during clinical trials.

A potential differentiating factor between delivering surveys via smart phone and other electronic modes of delivery is the perceived advantage of being able to conveniently complete survey questionnaires at any time and any location. This could help address certain limitations of the quantitative survey method such as recall bias. Furthermore, the portability, connectivity and ubiquity of smartphones may reduce the amount of training or instructions required for users to complete a survey questionnaire on a smartphone. For researchers, this type of survey delivery method may offer the benefits of a wider target audience and reduce research implementation costs. The e-PRO app is designed to further facilitate the delivery of PRO instruments in a convenient manner to participants. Through its computing capability, and user-friendly interface, the e-PRO app can collect data and implement complex scoring requirements, thus supporting the delivery of self-administered survey questionnaires. The goal of this two-arm randomized controlled pilot is to explore the usability and satisfaction with a novel e-PRO app.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants over the age of 18-65 years as assessed by the Self-Rated Health Measure.
* Fluency in English language to be able to read, understand study procedures and complete surveys administered during the study.
* Willing to travel to the downtown Boston area to participate in up to two study visits.
* Willing to participate in the research study and sign informed consent.

Exclusion Criteria:

* Participants with a "fair" or "poor" rating on the Self-Rated Health Measure.
* Participants with EU citizenship or permanent residency
* Participants with severe cognitive, vision, hearing, or speech problems that may prevent them from answering surveys
* Participants with serious psychiatric conditions (moderate or major depressive disorder that may impair their ability to complete surveys
* Participants with any terminal illness (e.g. cancers)
* Patients with implantable devices, pacemakers or body worn electronic medical devices

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Usability of e-PRO vs. emailed link: survey | At close-out
  A survey will be administered to compare groups on their experiences with the survey-method administration (Investigator developed survey). The following components will be taken into account: acceptability-- participant satisfaction with various aspects of the solution (e.g. content, complexity, comfort, delivery, and credibility). Adoption-- participants' intention to try; perceived barriers and facilitators for uptake. Appropriateness-- participant's perceived relevance to need; suitability to daily patient workflow. Feasibility-- suitability for using daily, weekly etc. This survey is not a scored survey.

SECONDARY OUTCOMES:
Survey response rate e-PRO vs emailed link | At close-out
  Response rate will be tracked on a weekly basis from the e-PRO system and the REDCap embedded email link to compare response rate between the control and intervention group. The AAOPR (2006) recommendation for RR formula will be used to calculate the RR. This is the number of completed surveys (completed and partially completed) divided by the number of completed surveys (completed and partially completed) plus the number of all non-completed surveys (sent to a potential participant but not completed because of incorrect e-mail address, incorrect mailing address, or other reasons).

CONTACTS AND LOCATIONS:
Overall Officials: Ramya S Palacholla, MD, MPH, Principal Investigator — Partners HealthCare
Locations (1):
- Partners Healthcare, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.